CLINICAL TRIAL: NCT07203573
Title: Prognostic Value of the C-Reactive Protein-Albumin-Lymphocyte (CALLY) Index on Patients Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Prognostic Value of the CALLY Index in Patients Undergoing Primary PCI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Madona Samy Anis, doctor, Assiut University
Other Study IDs: CALLY Index in PPCI Patients
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Primary Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the relationship between the admission CALLY index and short-term adverse outcomes in STEMI patients undergoing PPCI. Specifically, it seeks to determine whether the CALLY index is associated with in-hospital and 30-day complications, including heart failure, arrhythmias, reinfarction, or death. Additionally, the study will assess the association between the CALLY index and procedural success, defined by post-intervention TIMI flow, as well as the complexity of coronary artery disease using the SYNTAX score.

DETAILED DESCRIPTION:
* ST-elevation myocardial infarction (STEMI) remains a leading cause of morbidity and mortality worldwide. Early risk stratification in patients undergoing primary percutaneous coronary intervention (PPCI) is crucial to predict adverse outcomes and optimize management.
* The C-reactive protein-albumin-lymphocyte (CALLY) index is an emerging biomarker combining inflammation, nutrition, and immune status. Previous studies have demonstrated associations between the CALLY index and long-term mortality in cardiovascular disease, elderly populations, and STEMI patients . However, most of these studies focus on long-term outcomes or utilize complex predictive models (e.g., machine learning), and there is limited research assessing the direct relationship between admission CALLY index and immediate procedural outcomes, such as PPCI success or short-term adverse events., Unlike previous studies that included retrospective data, large national databases, or machine learning prediction models, this study will focus on a short-term, real-time assessment of the CALLY index at admission and its immediate association with procedural outcomes and in-hospital adverse events

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

* Diagnosis of STEMI based on 4th universal definition of myocardial infarction
* Undergoing Primary PCI within guideline-recommended timeframes
* Provided informed consent to participate in the study

Exclusion Criteria:

* Active infection (as detected by baseline leukocytosis on admission), autoimmune or inflammatory disease affecting CRP, albumin, or lymphocyte counts
* Chronic liver disease or advanced malignancy
* Patients receiving immunosuppressive therapy
* Refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years) presenting with STEMI to the emergency department and receiving PPCI as the main management
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Short-term major adverse cardiac events (MACE) | Through hospital stay (up to 3 days) and at one-month follow-up post-intervention.
  Occurrence of MACE including heart failure, arrhythmias, reinfarction, cardiogenic shock, or death.

SECONDARY OUTCOMES:
Procedural success of PPCI | Immediately post-procedure
  Achievement of final TIMI 3 flow grade post-intervention without in-hospital complications.
Coronary artery disease complexity by SYNTAX score ( (Synergy Between PCI With Taxus and Cardiac Surgery score) | At the time of coronary angiography
  Assessment of the association between CALLY index at admission and coronary complexity determined by the SYNTAX (Synergy Between PCI With Taxus and Cardiac Surgery) score.
  The SYNTAX score ranges from 0 upwards, with scores categorized as 0-22 indicating low complexity and scores >22 indicating more complex coronary artery disease. Higher scores represent increased disease complexity.

REFERENCES:
- [Background] Kumar R, Shah JA, Solangi BA, Ammar A, Kumar M, Khan N, Sial JA, Saghir T, Qamar N, Karim M. The Burden of Short-term Major Adverse Cardiac Events and its Determinants after Emergency Percutaneous Coronary Revascularization: A Prospective Follow-up Study. J Saudi Heart Assoc. 2022 Jun 11;34(2):100-109. doi: 10.37616/2212-5043.1302. eCollection 2022. PMID 36237223
- [Background] Ridker PM, Hennekens CH, Buring JE, Rifai N. C-reactive protein and other markers of inflammation in the prediction of cardiovascular disease in women. N Engl J Med. 2000 Mar 23;342(12):836-43. doi: 10.1056/NEJM200003233421202. PMID 10733371
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Demir Y, Sevinc S. The Prognostic Value of C-Reactive Protein-Albumin-Lymphocyte (CALLY) Index in Predicting In-Hospital Mortality After Primary Percutaneous Coronary Intervention in Patients With ST-Elevation Myocardial Infarction (STEMI). Catheter Cardiovasc Interv. 2025 Aug;106(2):1111-1118. doi: 10.1002/ccd.31623. Epub 2025 Jun 2. PMID 40452651
- [Background] Ji H, Luo Z, Ye L, He Y, Hao M, Yang Y, Tao X, Tong G, Zhou L. Prognostic significance of C-reactive protein-albumin-lymphocyte (CALLY) index after primary percutaneous coronary intervention in patients with ST-segment elevation myocardial infarction. Int Immunopharmacol. 2024 Nov 15;141:112860. doi: 10.1016/j.intimp.2024.112860. Epub 2024 Aug 13. PMID 39142002
- [Background] Guven B, Deniz MF, Geylan NA, Kultursay B, Donmez A, Bulat Z, Gul OB, Kaya M, Oktay V. A novel indicator of all-cause mortality in acute coronary syndrome: the CALLY index. Biomark Med. 2025 Apr;19(8):287-294. doi: 10.1080/17520363.2025.2483159. Epub 2025 Mar 24. PMID 40125936
- [Background] Fedai H, Sariisik G, Toprak K, Tascanov MB, Efe MM, Arga Y, Doganogullari S, Gez S, Demirbag R. A Machine Learning Model for the Prediction of No-Reflow Phenomenon in Acute Myocardial Infarction Using the CALLY Index. Diagnostics (Basel). 2024 Dec 14;14(24):2813. doi: 10.3390/diagnostics14242813. PMID 39767174
- [Background] Luo L, Li M, Xi Y, Hu J, Hu W. C-reactive protein-albumin-lymphocyte index as a feasible nutrition-immunity-inflammation marker of the outcome of all-cause and cardiovascular mortality in elderly. Clin Nutr ESPEN. 2024 Oct;63:346-353. doi: 10.1016/j.clnesp.2024.06.054. Epub 2024 Jul 2. PMID 38985666
- [Background] Kelemen Z, Mai A, Kapros T, Feher A, Gyorgyey J, Waterborg JH, Dudits D. Transformation vector based on promoter and intron sequences of a replacement histone H3 gene. A tool for high, constitutive gene expression in plants. Transgenic Res. 2002 Feb;11(1):69-72. doi: 10.1023/a:1013923826979. PMID 11874105